CLINICAL TRIAL: NCT04970212
Title: Pivotal Clinical Study to Establish the Safety and Effectiveness of the Use of BioTraceIO Lite for Assessment of Tissue Damage Following Liver Tissue Ablation Procedures
Brief Title: Safety and Effectiveness of BioTraceIO Lite for Tissue Damage Assessment Following Liver Tissue Ablation Procedures
Status: Completed | Type: Observational
Sponsor: Techsomed Medical Technologies LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CL000012
Record Dates: First submitted 2021-07-05; First posted 2021-07-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Hepatocellular; Metastatic Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Arm: Subjects will receive your standard liver ablation procedure, including ultrasound images. Data will be collected from the standard liver ablation procedure, including imaging. Subjects will receive a CT scan within 24 hours after the liver ablation procedure. There will then be an analysis of ultrasound images and research CT scan.
  Interventions: Device: BioTraceIO Lite

INTERVENTIONS:
Device: BioTraceIO Lite — The BioTraceIO software will analyze the ultrasound images, and provide the physician with an estimated tissue damage map.

SUMMARY:
Clinical study planned to demonstrate that the BioTraceIO Lite, available post-procedure, is effective at estimating the area of tissue damage as measured on 24-hour post-procedure (T=24hrs) CECT scan and that it is safe, based on an assessment of device-related Adverse Events.

Multi-center (up to 6 investigational sites) prospective single-arm clinical investigation 50 evaluable subjects total stratified by cancer type (primary hepatocellular carcinoma vs. secondary liver metastases).

DETAILED DESCRIPTION:
Clinical study planned to demonstrate that the BioTraceIO Lite, available post-procedure, is effective at estimating the area of tissue damage as measured on 24-hour post-procedure (T=24hrs) contrast-enhanced CT scan and that it is safe, based on an assessment of device-related Adverse Events.

BioTraceIO Lite is intended to provide physicians with adjunctive information in their clinical assessment of tissue damage created by liver tissue ablation, as part of their overall post-procedure clinical assessment.

Multi-center (up to 6 investigational sites) prospective single-arm clinical investigation 50 evaluable subjects total stratified by cancer type (primary hepatocellular carcinoma vs. secondary liver metastases).

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled and indicated for standard-of-care liver tissue ablation for either hepatocellular carcinoma (HCC) or metastatic liver tumor(s) using either RF or MW energy.
2. At least 21 years of age
3. Single tumor, or multiple tumors only if the distance between the ablated tumor and all other tumors allows for distinct separation between the necrotic zones (minimum of 1cm), based on the physician's discretion.
4. Distance between the tumor and the edge of any previous necrotic zones allows for distinct separation between the necrotic zones (minimum of 1cm), based on the physician's discretion.
5. Single ablation, using a single ablation needle, per tumor.
6. Able and willing to give informed consent.

Exclusion Criteria:

1. Liver tumor that cannot be ablated with a single ablation needle, according to the investigator's clinical opinion.
2. Subject cannot tolerate/undergo contrast-enhanced CT.
3. Planned ablation includes adjunctive means other than RF or MW energy (e.g., ethanol, hepatic artery embolization, etc.) or overlapping ablations using a single ablation needle.
4. Ablation area cannot be visualized continuously using ultrasound throughout the entire ablation procedure.
5. Pregnant or lactating
6. Currently participating in another clinical trial of an unapproved investigational device or drug that has not concluded the follow-up period.
7. Unable or unwilling to give informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been scheduled to have a liver ablation as part of their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-09-24 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Events | 1 year
  Incidence and severity of device-related adverse events (including serious adverse events (SAE)) occurring between the beginning of the liver tissue ablation procedure and the completion of the T=24hrs contrast-enhanced computed tomography (CECT) scan. There is no comparator for this endpoint.
Effectiveness - DICE | 1 year
  Paired comparison of the DICE similarity coefficient, assessed between BioTraceIO Lite, as measured at end of ablation procedure (T=0) and the tissue damage area based on 24-hours post-procedure CECT (T=24), and the DICE similarity coefficient, assessed between the tissue damage area based on immediately post-procedure CECT (T=0) and the tissue damage area based on 24-hours post-procedure CECT (T=24).

SECONDARY OUTCOMES:
Sensitivity | 1 year
  Sensitivity of the BioTraceIO Lite at T=0 compared to CECT at T=24hrs.
Precision | 1 year
  Precision of the BioTraceIO Lite at T=0 compared to CECT at T=24hrs.
Questionnaire - Effect of BioTraceIO | 1 year
  The proportion of subjects in whom the treating physician indicates that, if the BioTraceIO Lite results had been available for use in patient management, it would have impacted their follow-up plan for patient management, compared to the CECT alone.
Difference between T=0 and T=24hrs CECT tissue damage | 1 year
  Difference in percentage between tissue damage volume as visualized at T=0 contrast-enhanced computed tomography (CECT) versus tissue damage volume as visualized at T=24hrs CECT.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Stanford Medicine, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University Hospitals Cleveland, Cleveland, Ohio
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No